CLINICAL TRIAL: NCT04022174
Title: Effects of Action Observation and Motor Imagery on Orofacial Sensorimotor Variables
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Autonoma de Madrid (Other)
Responsible Party: Principal Investigator, Roy La Touche Arbizu, Principal Investigator, Universidad Autonoma de Madrid
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: uammadrid10
Record Dates: First submitted 2019-07-08; First posted 2019-07-16 (Actual); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Pain
Keywords: Motor Imagery; Action observation
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moderate dosage training (Experimental)
  Interventions: Behavioral: Moderate dosage training of action Observation and Motor imagery; Behavioral: Moderate dosage orofacial exercises
- Intensive dosage training (Experimental)
  Interventions: Behavioral: Intensive dosage training of action observation and motor imagery; Biological: Intensive dosage orofacial exercises

INTERVENTIONS:
Behavioral: Moderate dosage training of action Observation and Motor imagery — Motor imagery and action observation of orofacial exercises with moderate dosage
  Arms: Moderate dosage training
Behavioral: Intensive dosage training of action observation and motor imagery — Motor imagery and action observation of the orofacial exercises with intensive dosage
  Arms: Intensive dosage training
Biological: Intensive dosage orofacial exercises — Orofacial exercises with high intensity
  Arms: Intensive dosage training
Behavioral: Moderate dosage orofacial exercises — Orofacial exercises with moderate intensity
  Arms: Moderate dosage training

SUMMARY:
The main objective of the present study was to evaluate the effects of different dosages of action observation (AO) and motor imagery (MI) combined with an orofacial exercise program on pain pressure thresholds, lingual endurance and perceived exertion in asymptomatic subjects.

ELIGIBILITY:
Inclusion Criteria:

1. healthy individuals with no pain
2. aged between 18 and 65 years
3. subjects with correct masticatory function and labial and lingual mobility

Exclusion Criteria:

1. individuals who presented systemic, cardiorespiratory, central nervous system or rheumatic diseases, or those who presented any musculoskeletal or craniocervical pathology
2. underage individuals
3. individuals with orofacial pain or temporomandibular disorders at the time of the study
4. subjects' complaint of toothache or tenderness to percussion.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-07-12 (Estimated); Primary Completion 2019-08-12 (Estimated); Study Completion 2019-08-15 (Estimated)

PRIMARY OUTCOMES:
Pain pressure thresholds (PPTs) | Change from baseline and immediately post-intervention
  PPT is defined as the minimal amount of pressure where a sense of pressure first changes to pain. The mechanical pressure algometer (Force Ten TM FDX Digital Force Gage) used in this study consisted of a round rubber disk (area, 1 cm2) attached to a pressure (force) gauge. The gauge displays values in kilograms but, because the surface of the rubber tip is 1 cm2, the readings are expressed in kg/cm2. The range of values of the pressure algometer is 0 to 10 kg, with 0.1-kg divisions. The pressure was applied at a rate of 0.31 kg/second (Chesterton et al. 2007).
Lingual muscle endurance | Change from baseline and immediately post-intervention
  Lingual muscle endurance is assessed using the Iowa Oral Performance Instrument (IOPI) (Adams et al. 2015). The measurement of muscular endurance was carried out by placing a plastic bulb with oblong air content on the hard palate, posterior to the central incisor teeth. The participants were asked to elevate the lingual (through anterior and posterior lingual region) to press the instrument with the maximum possible force for 3 seconds, while monitoring the force exerted, quantified in Newtons Adams et al. (2015) found moderate to strong reliability for anterior (ICC: 0.58-0.77) and posterior (ICC 0.77-0.84) tongue strength.
Perceived exertion | Change from baseline and immediately post-intervention
  The Borg scale of perceived effort measures the entire range of effort that the individual perceives when exercising. This scale gives criteria to make adjustments to the intensity of exercise, that is. To the workload, and thus predict and dictate the different intensities of exercise in sports and in medical rehabilitation (BORG, 1982). It can also be used in athletics, astronautics, industry and military environments, as well as in everyday situations. The concept of perceived effort is a subjective evaluation that indicates the subject's opinion regarding the intensity of the work carried out (MORGAN, 1973). The subject doing the exercise must designate a number, from 1 to 20, to represent the subjective sensation of the amount of work performed and higher values represent more perceived exertion

CONTACTS AND LOCATIONS:
Locations (1):
- CSEU La Salle, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No